CLINICAL TRIAL: NCT03241082
Title: Use of Bedside Ultrasound to Assess Neonatal Body Composition in the Neonatal Intensive Care Unit
Brief Title: Ultrasound Assessment of BC in the NICU
Status: Active, not recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: PEDS-2017-25699
Record Dates: First submitted 2017-07-28; First posted 2017-08-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Premature Infant
MeSH Terms: conditions — Premature Birth | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ultrasound — validation of portable ultrasound to measure body composition

SUMMARY:
The overall objective of the proposal is to evaluate the ability of ultrasound to predict and routinely (weekly) monitor changes in the body composition of healthy preterm infants in the neonatal intensive care unit (NICU) in response to nutritional intake. The investigators hypothesize that ultrasound is an accurate method to routinely monitor the quality of weight gain and assess the adequacy of nutritional provision for premature infants in the neonatal intensive care unit.

The investigators will address the hypothesis in the following Specific Aims:

Specific Aim 1: Validate ultrasound as a method to measure whole body fat mass and fat free mass in healthy, premature infants. Body composition will be assessed using ultrasound measurements and the validated method of air displacement plethysmography (ADP). Stable isotope dilution techniques will be used in a subset of our population as a secondary source of validation.

Specific Aim 2: Determine whether ultrasound measurements can detect clinically relevant (weekly) changes in body composition in healthy premature infants. Ultrasound will be used to obtain serial (weekly) measurements of muscle and adipose tissue thickness (triceps, abdomen, quadriceps) until discharge in healthy, premature infants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, premature infants 25-34+6 weeks gestational age at birth
* Admitted to the University of Minnesota Masonic Children's Hospital NICU
* Stable on room air or can be removed from respiratory support for 5 minutes
* Written or verbal (telephone) informed consent can be secured from a parent within 1 week of admission to the NICU

Exclusion Criteria:

-Require medical support preventing ADP measurements

Ages: 25 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants admitted to the University of Minnesota NICU under the care of the PI and/or her colleagues.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Whole-body measurements of body composition | Up to 6 weeks
  Measurement of whole body fat mass and fat-free mass via air displacement plethysmography and stable isotope dilution.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Ramel, MD, Principal Investigator — University of Minnesota Department of Pediatrics
Locations (1):
- University of Minnesota Masonic Children's Hospital, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided